CLINICAL TRIAL: NCT05889130
Title: What Is the Optimal Timing for Intradialytic Resistance Exercise? A Randomized Controlled Trial
Brief Title: Optimal Timing for Resistance Exercise in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Ömer Bingölbali, Lecturer, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-86766
Record Dates: First submitted 2023-05-16; First posted 2023-06-05 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hemodialysis
Keywords: Hemodialysis; Resistant exercise; Blood Presure; Physical Performance; Quality of Life

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- first two hours of exercise group (Active Comparator): This is the group that will do resistance exercise in the first two hours of the hemodialysis session.
  Interventions: Other: Resistant Exercise
- last two hours of exercise group (Active Comparator): This is the group that will do resistance exercise in the last two hours of the hemodialysis session.
  Interventions: Other: Resistant Exercise

INTERVENTIONS:
Other: Resistant Exercise — The exercises were planned to be performed in 3 sets, 10 repetitions in each set, with 3 minutes rest between sets. Before starting the main exercises, it was planned to do 1 set of the same exercises without weight as a warm-up and cool-down exercise.
  Exercises were planned as lower extremity hip abduction, adduction, flexion and extension, straight leg raise, terminal knee extension, ankle flexion and bridge exercises. During the exercises, it was planned to be combined with breathing, paying attention to respiratory control.

SUMMARY:
The study consists of two groups doing resistance exercise for the first and last two hours of the HD session. The investigators are planning to form the sample size of exercise training from 40 participants, which the investigators determined according to the power analysis the investigators have done based on the blood pressure outcome criterion. Participants who meet the inclusion criteria the investigators have set will be divided into two groups. A resistance exercise training will be given three days a week for eight weeks, with a total of 24 sessions. The number of IRCAs occurring in both groups and blood pressure values to be measured at the beginning and end of the HD session will be checked, and both parameters will be compared between the groups before and after the treatment after 8 weeks of training. Thus, the investigators aim to show how the time factor has an effect on blood pressure. In addition, muscle strength, physical performance and quality of life of participants before and after resistance exercise will be evaluated and compared between groups. The participants' blood pressure will be evaluated with a conventional cuffed sphygmomanometer, muscle strength, digital hand dynamometer, physical performance, Short Physical Performance Battery and Timed Up and Go Test, and their quality of life will be evaluated with the Kidney Disease Quality of Life-36 (KDQOL-36) quality of life questionnaire. In exercise training, sandbags will be used as resistance. In our study, which the investigators planned as a randomized controlled trial, stratified randomization method will be used to distribute the gender factor homogeneously in both groups.

DETAILED DESCRIPTION:
Purpose and Objective: The aim of our study is to examine the effect of intradialytic (IR) resistance exercise time on blood pressure, physical performance and quality of life in hemodialysis (HD) patients. With this study we are planning to do, we aim to help HD patients regulate their blood pressure values and increase their muscle strength so that they can be more independent in their daily living activities and thus improve their quality of life.

Original Value: HD is the reorganization of the fluid and solute content of the blood taken from the patient by means of a membrane and with the help of a machine. The treatment requirements of HD patients (the HD session is usually applied two or three days a week and each application takes about 4 hours, as well as the plasma withdrawal from the body during HD) and long-term immobilization usually cause low blood pressure. This may cause some patients to have an intradialytic hypotensive attack (IDHA) due to the excessive decrease in blood pressure during HD. IDHA, on the other hand, is associated with severe abdominal pain, nausea, vomiting, dizziness, blackout, muscle cramps, with a decrease in systolic blood pressure of more than 20 mmHg compared to the predialysis (pre-dialysis) value or a decrease in mean systolic pressure of more than 10 mmHg from the predialysis value. It is defined as the coexistence of symptoms such as cramps and severe anxiety.

It is a known fact that regular exercises have a blood pressure lowering effect in the chronic period, and it is observed that exercises performed regardless of type (aerobic, resistant or combined) increase blood pressure in the acute period. Because blood flow is restricted due to the increase in pressure in the muscle during exercise, metabaroreceptors and mechanoreceptors in the active muscle stimulate the cardiovascular center in the medulla, and both systolic and diastolic pressure increase in order to exclude intramuscular pressure and provide perfusion. This is a response of the body to exercise and occurs as a result of normal physiological mechanisms.

Due to theoretical concerns that the exercise applied in the last two hours of the HD session may exacerbate hemodynamic instability, it is generally recommended to exercise in the first two hours of HD. However, there is also evidence showing that exercise can be done in the last two hours of the HD session. The increase in these evidences, especially in recent years, reveals that there is a need for studies on the effectiveness and reliability of IR exercise application time. The tendency of the blood pressure to drop more in the last half of the HD session (due to the increase in the amount of plasma withdrawn from the patients as time progresses) suggests that an exercise program that can be given in these minutes may provide a significant benefit to the patients, considering the acute blood pressure-raising effect.

From another point of view, studies show that resistance exercises (because it increases intramuscular pressure more) increase blood pressure more in the acute period than aerobic exercises. There are limited studies comparing the effects of aerobic and resistance exercises on blood pressure in HD patients. Limited existing studies have also revealed that resistance exercise raises blood pressure more than aerobic exercise in the acute period in HD patients. Therefore, it is thought that it would be more beneficial to include resistant exercises in the exercise program to be given to the patients in the last two hours.

However, many studies have proven that resistance exercises have a greater muscle strengthening effect when compared to aerobic exercises. It is known that the immobilization that HD patients are exposed to due to the long frequency and duration of dialysis sessions causes significant decreases in muscle strength. Therefore, it is expected that one of the main problems HD patients suffer from is falling, and there are studies supporting this situation. When all these points are evaluated, it is seen that resistance exercises are in a strategic position in HD patients. Therefore, considering the curative effect of muscle strengthening on physical performance parameters, it becomes important again that resistant exercises should be applied in HD patients. In addition, despite the limited range of motion of patients during HD, exercise therapy is not effective. It is extremely important that lay is a feasible treatment. However, since exercise therapy is relatively simple, easily applicable, non-invasive, and low-cost compared to other treatments, and also allows the patient to actively participate in his own treatment, it can also provide a useful self-management understanding in this sense by creating the perception that the patient is responsible for his own health. In addition, we think that the application of exercise therapy in HD units in our country will also support its spread, thanks to the effects we have mentioned above.

Method: Our study consists of two groups doing resistance exercise for the first and last two hours of the HD session. We are planning to form the sample size of exercise training from 40 patients, which we determined according to the power analysis we have done based on the blood pressure outcome criterion. Patients who meet the inclusion criteria we have set will be divided into two groups. A resistance exercise training will be given three days a week for eight weeks, with a total of 24 sessions. The number of IRCAs occurring in both groups and blood pressure values to be measured at the beginning and end of the HD session will be checked, and both parameters will be compared between the groups before and after the treatment after 8 weeks of training. Thus, we aim to show how the time factor has an effect on blood pressure. In addition, muscle strength, physical performance and quality of life of patients before and after resistance exercise will be evaluated and compared between groups. The patients' blood pressure will be evaluated with a conventional cuffed sphygmomanometer, muscle strength, digital hand dynamometer, physical performance, Short Physical Performance Battery and Timed Up and Go Test, and their quality of life will be evaluated with the Kidney Disease Quality of Life-36 (KDQOL-36) quality of life questionnaire. In exercise training, sandbags will be used as resistance. In our study, which we planned as a randomized controlled trial, stratified randomization method will be used to distribute the gender factor homogeneously in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Have been on HD treatment for at least 6 months
* To be receiving HD treatment for 4 hours 3 days a week
* 18 to 90 years old

Exclusion Criteria:

* Having angina pectoris or uncontrolled arrhythmia and uncontrolled hypertension
* Having communication or cognitive problems at a level that cannot fulfill the requirements of the tests
* Having an orthopedic problem that cannot do the exercise
* Have upcoming travel or kidney transplant plans
* Having an intradialytic hypotensive attack in 3 consecutive sessions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-05-13 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
systolic and diastolic blood pressure will be measured | Change from baseline and 8 weeks systolic and diastolic blood pressure

SECONDARY OUTCOMES:
The Short Physical Performance Battery Scale | baseline and 8 weeks
  The Short Physical Performance Battery (SPPB) is widely used to reduce the body and functional performance of the elderly living in the community. SPPB consists of 3 objective tests evaluating lower body structures. These; It is a 4 meter walking, standing up and standing balance test. A summary score of 5 levels (0-4) was assigned for each test. A score of zero indicates "Failure to fulfill". Participants included in the category of "not able to perform": 1- Those who tried to do the activity but could not do the activity, 2- The interviewer or the subject felt insecure, 3- Those who could not do the activity due to other health reasons (eg, too ill, too much follow-up monitoring). Scores of 1-4 obtained by the subjects show the progressive performance required to fulfill the test according to the times. The durations of the functions performed by the patients are recorded using a stopwatch.
Kidney Disease Quality of Life-36 | baseline and 8 weeks
  Quality of Life

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Mus Alparslan University, Muş, Güzeltepe District
  - Marmara University, Istanbul

IPD SHARING:
Plan to Share IPD: No